CLINICAL TRIAL: NCT06009432
Title: Efficacy of Proprioceptive Neuromuscular Facilitation Exercise Program Versus Usual Care in Patients With Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Efficacy of Proprioceptive Neuromuscular Facilitation Exercise Program in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kalça artroplasti pnf rkç
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hip Arthroplasty
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In addition to the program given to the control group, the study group will be given proprioceptive neuromuscular facilitation exercise as previously described (Smedes et. al., 2021). These applications will be applied to the patients for 8 weeks, 2 days a week in the clinical environment after the initial evaluation. In addition, both groups will be told that they can contact the researcher when requested.
  Interventions: Other: Rehabilitation
- Control Group (Active Comparator): The control group will receive the usual post-operative care of stretching lower extremity strengthening balance exercises activities of daily living recommendations.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — The control group will receive the usual post-operative care of stretching, lower extremity strengthening, balance exercises, activities of daily living recommendations. The study group will be given proprioceptive neuromuscular facilitation exercise in addition to the program given to the control group.

SUMMARY:
This study was planned to investigate the effectiveness of usual care and additional proprioceptive neuromuscular facilitation exercise program in patients undergoing total hip arthroplasty surgery. It is aimed to evaluate pain intensity, disability level, proprioception, kinesiophobia, balance and functional status of the patients. The study will be conducted with volunteer patients who are followed up by the Orthopedics and Traumatology outpatient clinic of Fethiye State Hospital and who have undergone total hip arthroplasty surgery. The evaluations will be performed in the Orthopedics and Traumatology outpatient clinic of Fethiye State Hospital. It is aimed to evaluate at least 42 patients for the study. The first evaluation will be performed 6 weeks post-operatively and the second evaluation will be performed 2 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone unilateral total hip arthroplasty surgery and being 6 weeks postoperative
* Participate in all necessary follow-up assessments
* 60 years of age or older
* Understand simple commands
* Signing the consent form

Exclusion Criteria:

* A previous history of total hip arthroplasty
* Presence of revision surgery
* Presence of severe osteoarthritis in the contralateral hip
* Severe acute metabolic neuromuscular and cardiovascular diseases
* Severe obesity (bki>35)
* Presence of malignancy
* Have any other orthopedic or neurological problem that may affect treatment and assessments
* Situations that prevent communication
* Lack of cooperation during the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from Baseline VAS at 8 weeks
  On a 10 cm straight line or numeric scale, the patient is asked to mark the pain they feel (0: no pain, 10: excruciating pain).
Western-Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change from Baseline WOMAC at 8 weeks
  Functionality level in the patient group with knee OA was measured using WOMAC. WOMAC consists of 3 main headings: pain intensity, stiffness and physical function. The individuals included in the study are asked to score each item between 0 (no pain, stiffness, difficulty) and 5 (very severe pain, stiffness, difficulty). The total score ranges from 0 (no disability) to 96 (complete disability).
3 Meter Backward Walk Test (3MBWT) | Change from Baseline 3MBWT at 8 weeks
  A distance of 3 meters is measured and marked. Children are asked to walk backwards safely when the signal is given and stop when they reach the marked point. They are allowed to look behind them if necessary. Measurements are repeated 3 times and the average time is recorded.
One Leg Standing Test (OLST) | Change from Baseline OLST at 8 weeks
  The subject is tested standing on one leg using the right and left legs respectively. The test is repeated on a hard surface with eyes open and closed. The subject is asked to place both hands on the hips and look at a target on the wall at eye level at a distance of 1 meter. The subject is asked to stand with one leg in a 90 degree flexion position and the other leg in a standing position. A stopwatch is used to record the time the subject can maintain the test position. If the subject can hold the position for more than 30 seconds, the test is terminated and the elapsed time is recorded.
Five Times Sit to Stand Test (5TSST) | Change from Baseline 5TSST at 8 weeks
  A chair without armrests, with a 28.5 cm deep seat and backrest and adjustable height is used for the tests. Subjects start in a seated position, with their arms in the desired position and their backs against the chair backrest. The following verbal instructions are given: "Please stand up and sit down 5 times as quickly as possible. Straighten your knees when standing up and lean your back against the backrest when sitting down." Timing with the digital stopwatch is started manually with the instruction "Start" and stopped when the subject's back touches the backrest after the fifth standing up.
Fear-Avoidance Beliefs Questionnaire (FABQ) | Change from Baseline FABQ at 8 weeks
  The FABQ consists of 16 items and is divided into 2 subscales. The items are scored on a 7-point Likert scale (from strongly disagree to strongly agree). The score of each subscale is used independently. Higher scores represent more fear avoidance beliefs.
Falls Efficacy Scale International (FES-I) | Change from Baseline FES-I at 8 weeks
  The FES-I is a self-report questionnaire, providing information on level of concern about falls during activities of daily living. The questionnaire contains 16 items scored on a four-point scale (1 = not at all concerned to 4 = very concerned) providing a total score ranging from 16 (absence of concern) to 64 (extreme concern).
Hip joint proprioception measurement | Change from Baseline proprioception measurement at 8 weeks
  Patients were placed in a supine position and blindfolded to eliminate visual cues. The test started at neutral position (0°) and patient actively fexed the hip toward the fexion target position of 45°, which was indicated by a mechanical obstruction. After holding that position for 5 s, patient focused and remembered the angle, and brought the joint actively back to the neutral starting position. Then, patient was asked to actively reproduce the target position without the mechanical obstruction and hold at where he/she felt it was the just position. Five repetitions were performed for each leg and "absolute angular error" values were obtained from the start and stop angles.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özden, PhD, Study Director — Muğla Sıtkı Koçman University
Locations (1):
- Muğla, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No